CLINICAL TRIAL: NCT02576483
Title: An Evaluation of Quality of Vision and Quality of Life With LASIK, SMILE and PRK Surgery in Physicians
Brief Title: An Evaluation of LASIK, SMILE and PRK Surgery in Physicians
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Principal Investigator, Stanford University
Other Study IDs: 34287
Record Dates: First submitted 2015-09-28; First posted 2015-10-15 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Nearsightedness; Farsightedness; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Questionnaire (QoV questionnaire) — Quality of vision and quality of life questionnaire

SUMMARY:
The principle investigator is evaluating self-reported quality of vision and quality of life in physicians undergoing LASIK, SMILE and PRK surgery.

DETAILED DESCRIPTION:
The participants will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the participant from the study, then the investigator will inform the participant and make an appropriate referral. This is standard practice for laser in situ keratomileusis (LASIK) surgery, small incision lenticule extraction (SMILE) and photorefractive keratectomy (PRK) surgery.

If the participant is deemed appropriate for the study after a comprehensive examination including computerized videokeratography, then the participant can be enrolled. These exams are also standard practice for LASIK, SMILE and PRK surgery.

The Quality of Vision (QoV) Questionnaire will be administered following the pre-operative visit during which participants are enrolled and then at the three-month and twelve-month post- op visits before the participants are seen by the principle investigator. The questionnaire is the study intervention.

The participant will undergo bilateral simultaneous LASIK eye surgery, SMILE or PRK surgery. The participants will be seen pre-operatively, on the day of surgery, post op day one, one month, three months, and twelve-months as part of the study. Participants may also be seen more frequently if required from a medical standpoint. The participant will receive topical antibiotics in each eye for one week following the procedure. LASIK treated eyes will receive pred forte 1% ophthalmic drops for one week to four weeks after treatment. All of this is within the usual and customary standard of care for the treatment of patients undergoing LASIK, SMILE and PRK surgery.

ELIGIBILITY:
Inclusion criteria.

* 21 years or older.
* A physician or medical student.
* Have the ability to give informed consent.
* Speak and read English fluently.
* Have not previously had any form of refractive surgery, including prior LASIK or cataract surgery.
* May benefit from increased spectacle independence.
* Have been determined to be a good candidate for the LASIK, SMILE or PRK procedure based on the investigator's assessment of medical and ophthalmic health, general cognitive function, and physical and social limitations.
* Have a treatment target of bilateral emmetropia.
* Express willingness and potential ability to return for all follow-up examinations through the 12-month follow-up exam under the care of the treating investigator.
* Are not enrolled in any other research study.

Exclusion criteria.

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectatic eye disorders.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physicians with refractive errors
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported quality of vision and quality of life questionnaire | Twleve months

SECONDARY OUTCOMES:
Predictability (Percentage of eyes within 0.25, +/- 0.50 and +/- 1.00 diopters of the intended correction | Preoperatively, one, three, six and twelve months
Changes in CDVA (Corrected distance visual acuity) | Preoperatively, one, three, six and twelve months
Changes in low contrast acuity (5% and 25% contrast acuity) | Preoperatively, one, three, six and twelve months
Self-reported quality of life and quality of vision (QoV questionnaire) | Preoperatively, one, three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States